CLINICAL TRIAL: NCT02022046
Title: Methylation Biosignature in Childhood Chronic Kidney Disease: the Link Among Asymmetric Dimethylarginine, Homocysteine, and Cardiovascular Disease
Brief Title: Methylation Biosignature in Childhood Chronic Kidney Disease
Acronym: childhoodCKD
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Tain, You-Lin, MD, PhD, Chang Gung Memorial Hospital
Other Study IDs: 102-4131C
Record Dates: First submitted 2013-12-11; First posted 2013-12-27 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Chronic Kidney Disease; Cardiovascular Disease
Keywords: chronic kidney disease; cardiovascular disease; nitric oxide; homocysteine; asymmetric dimethylarginine; methylation
MeSH Terms: conditions — Renal Insufficiency, Chronic; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 2/study, control: Study group: children aged<18 years with chronic kidney disease Control group: children aged<18 years without chronic kidney disease Methylation biosignature, CKD staging, assessment of cardiovascular function, and traditional/uremia-related risk factors will be performed.
  Interventions: Other: Methylation biosignature

INTERVENTIONS:
Other: Methylation biosignature — Methylation biosignature, CKD staging, assessment of cardiovascular function, and traditional/uremia-related risk factors will be performed.

SUMMARY:
Chronic kidney disease (CKD) and end-stage renal disease are highly prevalent in Taiwan. Cardiovascular disease (CVD) is the most common cause of death in children with CKD. Nitric oxide (NO) deficiency links CKD and CVD. Asymmetric dimethylarginine (ADMA), a NO synthase inhibitor, its level is increased in kidney disease and cardiovascular disease and serves as a methylation biomarker.

In addition to ADMA, uremic environment, hyperhomocysteinemia (Hcy) and oxidative stress may affect DNA methylation. S-adenosylmethionine (SAM) is an important human methyl donor. S-adenosylhomocysteine (SAH) is demethylated product. Methylenetetrahydrofolate reductase (MTHFR), a folate metabolism enzyme can regulate methylation pathway.

The investigators intend to examine whether ADMA, SAM/SAH ratio, Hcy, and MTHFR gene methylation can serve as biosignature to predict CVD in children with CKD children.

ELIGIBILITY:
Inclusion Criteria:

* chronic kidney disease stage 1-4
* Volunteer

Exclusion Criteria:

* pregnancy
* renal transplant
* congenital heart disease
* not able to be adherent/complaint with study procedure
* not volunteer

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children aged <18 years visit pediatric nephrology clinic during study period
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2014-04; Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
change from baseline level of asymmetric dimethylarginine (ADMA) at 24 months | from the time of enrollment, every 6 months, up to 24 months
  at the time of enrollment, 6 months, 12 months, 18 months, and 24 months

SECONDARY OUTCOMES:
change from the baseline health-related quality of life at 24 months | from the time of enrollment, every 6 months, up to 24 months
  EQ-5D-Y instrument will be employed at the time of enrollment, 6 months, 12 months, 18 months, 24 months
change from the baseline ratio of SAM/SAH (S-adenosylmethionine /S-adenosylhomocysteine ) at 24 months | from the time of enrollment, every 6 months, up to 24 months
  at the time of enrollment, 6 months, 12 months, 18 months, 24 months
change from the baseline level of hyperhomocysteinemia (Hcy) at 24 months | from the time of enrollment, every 6 months, up to 24 months
  at the time of enrollment, 6 months, 12 months, 18 months, 24 months

CONTACTS AND LOCATIONS:
Overall Officials: You-Lin Tain, MD, PhD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan